CLINICAL TRIAL: NCT03255213
Title: Lingual Muscle Training in Late-Onset Pompe Disease (LOPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00077344
Record Dates: First submitted 2017-08-03; First posted 2017-08-21 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Glycogen Storage Disease
MeSH Terms: conditions — Glycogen Storage Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Late Onset Pompe Disease who have tongue weakness (Experimental)
  Interventions: Other: Lingual Muscle Training

INTERVENTIONS:
Other: Lingual Muscle Training — Lingual Muscle Training using the Iowa Oral Performance Instrument (OIPI) device

SUMMARY:
This study is being done to test the effects of Lingual Muscle Therapy (LMT) in patients with Late-Onset Pompe Disease (LOPD) who have tongue weakness. The results of this study will help design future research studies about LMT in LOPD.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 12 years
* Lingual weakness as measured by quantitative muscle testing (≤ 5% lower limit of normal for stratified age)
* Confirmed diagnosis of LOPD
* On enzyme replacement therapy for ≥ 26 weeks at pretest
* Able to follow directions for study participation
* Able to complete a home-based LMT regimen
* Access to reliable internet connection
* Access to use of electronic device that allows for FaceTime, Jabber, or WebEx use

Exclusion Criteria:

* Neurodegenerative conditions (e.g. stroke, dementia) or other serious neurologic condition that would prevent meaningful study participation as determined at the discretion of the principle investigator
* Any current or past history of seizures.
* Head and neck cancer or radiation treatment to head/neck
* Inability to tolerate IOPI device tongue bulb
* Inability to give legally effective consent
* Inability to read and understand English

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Safety of lingual muscle training | 13 weeks
  Safety measured by pain rating scale
Feasibility of lingual muscle training as measured by questionnaires | 13 weeks

SECONDARY OUTCOMES:
Change in lingual strength | baseline, 13 weeks
  Change from pre-test to post-test

CONTACTS AND LOCATIONS:
Overall Officials: Jones Harrison, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center and affiliated practices, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No